CLINICAL TRIAL: NCT02149953
Title: Determination Glycine Requirements During Healthy Pregnancy Using the Indicator Amino Acid Oxidation (IAAO) Technique
Brief Title: Determination of Glycine Requirement in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H14-00495; F13-04173 (Other Grant/Funding Number: Canadian Institute of Health Research)
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy
Keywords: Pregnancy; Glycine requirements; Indicator Amino Acid Oxidation (IAAO) method; Stable isotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glycine intake (Experimental): Dietary supplement: Glycine intake
  Interventions: Dietary Supplement: Glycine Intake

INTERVENTIONS:
Dietary Supplement: Glycine Intake — Oral consumption of eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.

SUMMARY:
It is important that pregnant women eat an adequate amount of protein to ensure healthy growth and development of the fetus. Amino acids are the building blocks of the body's protein. Glycine is an amino acid that can be made in the body, but under certain metabolic circumstances (e.g. pregnancy) the body's needs may be higher and thus glycine must be obtained from the diet. Currently, it is not known how much glycine may be needed from the diet during pregnancy. We plan to study dietary glycine requirements in healthy pregnant women, during early and late gestation. We will do this using a modern, safe and quick method.

DETAILED DESCRIPTION:
Purpose:

To determine the dietary glycine requirement in healthy pregnant women during mid (20 - 30 weeks) and late (31 - 40 weeks) gestation.

Hypothesis:

We hypothesize that there is a dietary requirement for glycine during pregnancy due to an increased metabolic demand. With increased glycine intake we hypothesize to observe an increase in protein synthesis, as measured by the indicator amino acid oxidation (IAAO) method.

Justification:

Inadequate protein intake during pregnancy may cause intrauterine growth restriction, which is associated with increased risk of chronic diseases later in life. Currently, the dietary intake recommendations for amino acids are greatly based on nitrogen balance studies of non-pregnant adults. There is little scientific information regarding dietary glycine needs during different stages of pregnancy, despite empirical evidence indicating gestational differences in protein metabolism.

Objectives:

The main objective of the current study is to determine the glycine requirement using the minimally invasive indicator amino acid oxidation (IAAO) method in healthy pregnant women. Our second objective is to compare the glycine requirement during mid (20-30 weeks gestation) and late (31 - 40 weeks gestation) stages of pregnancy.

Research methods:

We will recruit a minimum of 18 pregnant women who may take part in 2 study days in both gestational stages, for a total of 72 study days. Potential participants will meet us for a preliminary assessment where we will evaluate their eligibility to participate in the study. The preliminary study will take approximately 1 hr during which we will examine body composition (bioelectrical impedance, skin-fold measurements, height and weight), resting energy expenditure (indirect calorimetry), blood glucose (glucometer), and medical history (questionnaire). Fasted blood glucose above 6.7 mmol/L is indicative of gestational diabetes. Participants with fasted blood glucose concentrations above 6.7 mmol/L will be referred to follow-up with their primary health care provider (see letter to physician).

We will test the participants urine using a dipstick, to assess whether proteinurea is present. If there is an indication of proteinurea we will refer the participant to their primary physician (See letter to physician - Urine results).

We will collect a 3 day diet record to determine usual food intake and food preferences. Based on the 3 day food record we will prescribe a standardized diet two days prior to the study day to ensure protein intake of 1.5 g/kg/d and energy intake of 1.7 x resting energy.

During each study day, eligible participants will randomly receive 1 of 36 test glycine intakes during both mid and late pregnancy, ranging from 10 to 100 mg/kg/d. Each subject may participate in 2 study days between 20-30 weeks gestation and 2 study days between 31 - 40 weeks gestation, for a total of 4 study days. The test glycine intakes will contain a crystalline L-amino acid mixture based on the composition of egg protein, except for glycine. The test glycine intake will be administered in an experimental diet, along with enough non-protein energy to meet 1.7 x resting energy expenditure of each participant. The diet will be provided as 8 meals, each representing 1/12th of the participant's daily intake requirement. These meals will be provided over the course of an 8 hour study day. A stable isotope tracer will be added to the 5th - 8th meal. We will measure the rate of oxidation of this tracer in expired breath (F13CO2), and flux of this tracer by its enrichment in urine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women aged 20 - 40 yrs
* Singleton pregnancy
* Mid (20 - 30 weeks of gestation) or late stages of pregnancy (31 - 40 weeks of gestation).
* In good health (Free of chronic diseases/acute diseases, full range of physical mobility)

Exclusion Criteria:

* Women who are not pregnant
* Women who are pregnant with more than one child
* Women with history of spontaneous abortion, pre-term birth
* Women who are not in good health or have metabolic, neurologic or immune disorders including; preeclampsia/eclampsia, gestational diabetes, pregnancy-related anemia, pregnancy- related jaundice.
* Women who are substance dependent (i.e. alcohol, cigarette, illicit drugs)
* Women allergic to egg/ egg protein
* Women who have experienced severe nausea and vomiting throughout pregnancy
* Women who are claustrophobic

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
13 Carbon dioxide production | 8 hours
  Urine, breath and a single blood sample will be collected during the study to measure the rate of oxidation of tracer in expired breath and flux by enrichment in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen BF, Ennis MA, Dyer RA, Lim K, Elango R. Glycine, a Dispensable Amino Acid, Is Conditionally Indispensable in Late Stages of Human Pregnancy. J Nutr. 2021 Feb 1;151(2):361-369. doi: 10.1093/jn/nxaa263. PMID 32939556